CLINICAL TRIAL: NCT00253812
Title: Adenoma Detection Rate in Rectal Remnants of Familial Polyposis (FAP) Patients Using Standard (White Light), Auto-Fluorescence (AFI), Narrow Band Imaging (NBI) and Chromoscopic Endoscopy
Brief Title: Adenoma Detection Rate:NBI, AFI, Chromoscopic or Standard Endoscopy
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: London North West Healthcare NHS Trust (Other)
Allocation: Non-Randomized | Model: Crossover | Masking: Single | Purpose: Diagnostic
Other Study IDs: 05ADR-88
Record Dates: First submitted 2005-11-11; First posted 2005-11-15 (Estimated); Last update posted 2007-09-24 (Estimated); Status verified 2007-09

CONDITIONS: Familial Adenomatous Polyposis
Keywords: colonoscopy, sigmoidoscopy, chromoendoscopy, autofluorescence, narrow band imaging, colorectal cancer, polyp, adenoma,rectal remnant, FAP
MeSH Terms: conditions — Adenomatous Polyposis Coli; Colorectal Neoplasms; Polyps; Adenoma

INTERVENTIONS:
Procedure: flexible sigmoidoscopy

SUMMARY:
The purpose of this study is to establish whether new techniques that may make polyps (adenomas) stand out better from the background help increase the number of polyps visible at sigmoidoscopy (telescope test to look inside large bowel) compared to looking with standard sigmoidoscopy alone.

DETAILED DESCRIPTION:
Colorectal cancer is the second commonest cause of cancer death. In majority of cases it is preceeded by a precancerous lesion called an adenoma (commonly known as polyp). Detection and removal of adenomas has been shown to reduce the death rate from colorectal cancer. Despite of meticulous examination "a miss rate" for adenomas at colonoscopy ranges from 6-15% in back-to-back colonoscopy studies. The nature of the polyps, which as well as being pedunculated (cherry like) can also be flat, which makes it difficult to see and detect and may add to the"miss rate".

The factors that affect whether an endoscopist sees a polyp are not well studied. Polyp detection rates vary widely, even amongst experts. Techniques that highlight lesions advanced in recent years. Chromoendoscopy, spraying dye on the bowel lining, has been shown to help pick up more precancerous polyps in one of three studies in normal patients. Autofluorescence endoscopy (AFI) and narrow band imaging (NBI) use light filters to produce a false colour image of the bowel lining where polyps stand out. These techniques have been used with some success in the oesophagus and stomach but little work is available for the colon.

Patients with familial adenomatous polyposis (FAP) have many hundreds of bowel polyps due to a genetic defect and are at very high risk of colorectal cancer. Many of them have the majority of the large bowel removed with only lowest part of the large bowel, the rectum, left and joined to the small bowel. The remaining rectum can still have up to 50 polyps and is regularly surveilled with sigmoidoscopy to see if any large polyps have grown so they can be removed before they turn into cancer. Some of these polyps are small and flat.

We aim to see if using the new enhancement techniques we can detect more polyps in patients with FAP than with standard endoscopy.The patients will undergo flexible sigmoidoscopy as usual. This will then be repeated with the auto fluorescence feature of the endoscope activated, followed by a repeat with the narrow band feature activate. Then the lining of the bowel will be sprayed with blue dye (non-absorbed) and extra dye suctioned, the viewing process will be repeated the final time. This should take approx. 5 minutes. The videos from the procedures will be anonymised and randomised for viewing by another endoscopist.

ELIGIBILITY:
Inclusion Criteria:

* Patients with Familial adenomatous polyposis who have had ileo-rectal anastomosis and had 20 or less adenomas at previous surveillance examination

Exclusion Criteria:

* poor bowel preparation, unable or unwilling to give informed consent, under 18 years of age,those with more than 20 adenoma

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 60 (Estimated)
Dates: Start 2005-11

PRIMARY OUTCOMES:
The primary outcome measure will be the mean number of adenomas detected on the blinded video review for each endoscopy

SECONDARY OUTCOMES:
Adenoma detection rate for each of the modalities compared with each other.
Primary endoscopist adenoma count for each modality.

CONTACTS AND LOCATIONS:
Overall Officials: Brian Saunders, MD, FRCP, Study Director — Nort West London Hospitals NHS Trust - St Mark's Hospital
Locations (1):
- Norht West London Hospitals NHS Trust, London, Middlesex, United Kingdom